CLINICAL TRIAL: NCT00267540
Title: Adolescent Girls-Impact of Vitamin D on Bone Accretion Work Package 1 (Danish Part) of OPTIFORD (Towards A Strategy for Optimal Vitamin D Fortification)
Brief Title: The Effect of Vitamin D on Bone Accretion and Turn-Over in Young Girls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Seventh Framework Programme (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: QLK1-CT-2000-00623
Record Dates: First submitted 2005-12-20; First posted 2005-12-21 (Estimated); Last update posted 2008-01-30 (Estimated); Status verified 2008-01

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D; adolescent girls; bone accretion; bone turn over; vitamin D status; Vitamin D insufficiency in young girls
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol; Vitamins

INTERVENTIONS:
Behavioral: cholecalciferol (D3) (vitamin)

SUMMARY:
Objectives To evaluate the effect of increased vitamin D intake on vitamin D status, bone mass and bone turnover in young girls aged 12-13.

More specifically the effects on the following parameters will be assessed:

* Vitamin D metabolites.
* Parathyroid hormone.
* Bone turnover.
* Bone mineral accretion.
* Serum calcium and phosphate.
* Renal handling of calcium and phosphate.

DETAILED DESCRIPTION:
This work package will consist of a randomised double blind one-year vitamin D supplementation study. Primary effect parameter is change in bone mineral content and therefore study duration will be one year. A total of 225 subjects, 75 in each of the three groups: one control and two intervention groups, will be included Two dosages of supplementation will be used: 5 µg per day and 10 µg per day.

ELIGIBILITY:
Inclusion Criteria:

* Girls born in Denmark with Danish citizenship aged 10.0-11.0 years living in the municipals of Copenhagen and Frederiksberg

Exclusion Criteria:

* Any chronical disease with influence on bone mass or turnover
* Intake of drugs with influence on bone mass or turnover
* Intake of calcium or vitamin D other than the intervention

Ages: 10 Years to 11 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 225
Dates: Start 2001-01; Study Completion 2003-12

PRIMARY OUTCOMES:
Vitamin D level (status) measured as s-25 hydroxy vitamin D at baseline, after half a year and one year.
Bone accretion measured by DXA. Measurement at baseline and after one year.
Bone turnover measured at baseline, half a year and one year

CONTACTS AND LOCATIONS:
Overall Officials: Christian Mølgaard, MD, PhD, Principal Investigator — The Royal Veterinary and Agricultural University, Frederiksberg, Denmark
Locations (1):
- Department of Human Nutrition, The Royal Veterinary and Agricultural University, Frederiksberg, Denmark

REFERENCES:
- [Derived] Cashman KD, FitzGerald AP, Viljakainen HT, Jakobsen J, Michaelsen KF, Lamberg-Allardt C, Molgaard C. Estimation of the dietary requirement for vitamin D in healthy adolescent white girls. Am J Clin Nutr. 2011 Mar;93(3):549-55. doi: 10.3945/ajcn.110.006577. Epub 2011 Jan 26. PMID 21270380